CLINICAL TRIAL: NCT03409341
Title: Personalizing Immune Checkpoint Inhibitor Therapy for Solid Tumors
Brief Title: Personalizing Immune Checkpoint Inhibitor Therapy
Status: Withdrawn | Type: Observational
Why Stopped: No enrollment
Sponsor: Holy Cross Hospital, Maryland (Other)
Responsible Party: Sponsor
Other Study IDs: IRB# 2018-02
Record Dates: First submitted 2018-01-18; First posted 2018-01-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Lung Cancer Stage IV
MeSH Terms: conditions — Lung Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Peripheral blood samples will be used to evaluate immune cell anti-tumor response, and DNA sequence.
  2. A sample of tumor tissue excised for diagnostic biopsy will be used to evaluate tumor immunogenicity, tumor transcriptome, tumor infiltrating immune cells, and tumor DNA sequence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood and tumor tissue analysis, Clinical response. — DNA sequencing and functional testing of peripheral blood mononuclear cells. DNA and RNA sequencing and immune cell analysis of tumor. Clinical response at 12 months.

SUMMARY:
This prospective, observational study will evaluate whether vitro testing of tumor tissue and white blood cells from patients with lung cancer who are being treated with immune checkpoint inhibitors and other standard of care approaches, predicts clinical response to these agents.

DETAILED DESCRIPTION:
Overall Goal: The long-term goal of this study is to predict whether checkpoint inhibitors will be effective in individual patients with solid tumors.

Objectives: In this pilot study to be conducted in ten subjects with lung cancer who are to receive checkpoint inhibitors, we will use cellular and molecular techniques to characterize

* tumor immunogenicity
* anti-tumor T-cell response
* effect of checkpoint inhibitors on antigen presentation and T-cell response, and
* the tumor microenvironment

Planned enrollment:

• Ten subjects with lung cancer

Methods for Informed Consent:

Investigators will approach subjects for informed consent

ELIGIBILITY:
Inclusion Criteria:

* Subjects with lung cancer about to undergo diagnostic/excisional biopsy with the intent to receive therapy with immune checkpoint inhibitors
* Availability of fresh tumor tissue removed at excisional biopsy or diagnostic biopsy
* Informed consent

Exclusion Criteria:

• Lack of informed consent

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: • Ten subjects with lung cancer about to undergo diagnostic/excisional biopsy with the intent to receive therapy with immune checkpoint inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Anti-tumor immune response | 12 months
  Tumor antigen presentation and anti-tumor T-cell response

SECONDARY OUTCOMES:
Clinical response | 12 months for each subject
  Clinical response is defined as 50% or greater decrease of the sum of the products of two-dimensional measurements of lesions on imaging within the first year.
Tumor microenvironment | 24 months total study duration
  Tumor mutation burden from tumor genome landscape using DNA sequencing, tumor transcriptome with RNA sequencing, tumor infiltrating immune cells with flow cytometry

CONTACTS AND LOCATIONS:
Locations (1):
- Holy Cross Hospital, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing: The data generated in this study will be available to The Holy Cross Health Institutional Review Board, Inc., Investigators named in this protocol, and Officials of the FDA and HHS. Published information following completion of the study will be provided to study patients.
Supporting Information: CSR
Time Frame: 24 months
Access Criteria: Upon completion, published results will be provided to participants

REFERENCES:
- [Background] Sindhi R, Ashokkumar C, Higgs BW. Cellular alloresponses for rejection-risk assessment after pediatric transplantation. Curr Opin Organ Transplant. 2011 Oct;16(5):515-21. doi: 10.1097/MOT.0b013e32834a94e3. PMID 21844808
- [Background] Ashokkumar C, Talukdar A, Sun Q, Higgs BW, Janosky J, Wilson P, Mazariegos G, Jaffe R, Demetris A, Dobberstein J, Soltys K, Bond G, Thomson AW, Zeevi A, Sindhi R. Allospecific CD154+ T cells associate with rejection risk after pediatric liver transplantation. Am J Transplant. 2009 Jan;9(1):179-91. doi: 10.1111/j.1600-6143.2008.02459.x. Epub 2008 Oct 31. PMID 18976293
- [Background] Ningappa M, Ashokkumar C, Higgs BW, Sun Q, Jaffe R, Mazariegos G, Li D, Weeks DE, Subramaniam S, Ferrell R, Hakonarson H, Sindhi R. Enhanced B Cell Alloantigen Presentation and Its Epigenetic Dysregulation in Liver Transplant Rejection. Am J Transplant. 2016 Feb;16(2):497-508. doi: 10.1111/ajt.13509. Epub 2015 Dec 11. PMID 26663361
- [Background] Ranganathan S, Ningappa M, Ashokkumar C, Higgs BW, Min J, Sun Q, Schmitt L, Subramaniam S, Hakonarson H, Sindhi R. Loss of EGFR-ASAP1 signaling in metastatic and unresectable hepatoblastoma. Sci Rep. 2016 Dec 2;6:38347. doi: 10.1038/srep38347. PMID 27910913
- [Background] Vinayak R, Cruz RJ Jr, Ranganathan S, Mohanka R, Mazariegos G, Soltys K, Bond G, Tadros S, Humar A, Marsh JW, Selby RR, Reyes J, Sun Q, Haberman K, Sindhi R. Pediatric liver transplantation for hepatocellular cancer and rare liver malignancies: US multicenter and single-center experience (1981-2015). Liver Transpl. 2017 Dec;23(12):1577-1588. doi: 10.1002/lt.24847. PMID 28834194
- [Background] Cruz RJ Jr, Ranganathan S, Mazariegos G, Soltys K, Nayyar N, Sun Q, Bond G, Shaw PH, Haberman K, Krishnamurti L, Marsh JW, Humar A, Sindhi R. Analysis of national and single-center incidence and survival after liver transplantation for hepatoblastoma: new trends and future opportunities. Surgery. 2013 Feb;153(2):150-9. doi: 10.1016/j.surg.2012.11.006. PMID 23331862